CLINICAL TRIAL: NCT03205098
Title: Evaluation of Biological Markers of Mesenteric Ischemia During an Ultra-trail
Acronym: ISKETRAIL
Status: Completed | Type: Observational
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Other Study IDs: CHU-340; 2015-A00470-49 (Other: 2015-A00470-49)
Record Dates: First submitted 2017-06-21; First posted 2017-07-02 (Actual); Last update posted 2017-07-02 (Actual); Status verified 2017-06

CONDITIONS: Ultra-trail Participation
Keywords: biological markers; mesenteric ischemia; ultratrail
MeSH Terms: conditions — Mesenteric Ischemia | interventions — Hematologic Tests

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Runners: To assess the evolution of biological markers of mesenteric ischemia during ultratrail.
  Interventions: Biological: Blood analysis

INTERVENTIONS:
Biological: Blood analysis — Blood test of biological markers of mesenteric ischemia

SUMMARY:
To assess the evolution of biological markers of mesenteric ischemia during ultratrail.

DETAILED DESCRIPTION:
During physical exercise, increased sympathetic nervous system activity redistributes blood flow from splanchnic organs to working muscles. With prolonged duration and / or intensity, the splanchnic blood flow can be reduced by 80% or more. A severely reduced of splanchnic blood flow can frequently cause gastrointestinal ischemia. This ischemia associated with reduced vagal activity probably results in changes in motility and absorption.

High symptoms are reported in 40% of runners with reflux and heartburn in 15-20% of runners. The low symptoms have an incidence of about 70% in the long runs type ultra-trail.

Biological markers such as I-FABP have been shown to be useful in the diagnosis of mesenteric ischemia.

ELIGIBILITY:
Inclusion Criteria:

* Healthy Voluntary Subject
* Age > 18 years
* Written consent
* Subject affiliated to Social Security
* Medical certificate (mandatory to take part in the ultra-trail)

Exclusion Criteria:

* Refusal to participate
* Subject with legal protection (guardianship, trusteeship)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: participants or populations are selected based on predefined criteria
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2015-06-19 (Actual); Primary Completion 2015-06-30 (Actual); Study Completion 2016-09-30 (Actual)

PRIMARY OUTCOMES:
Assess biological markers of mesenteric ischemia (IFABP) | at day 1
  during ultratrail.

SECONDARY OUTCOMES:
Relationship between digestive symptoms and biological markers (IFABP). | at day 1

CONTACTS AND LOCATIONS:
Overall Officials: Sébastien PERBET, Principal Investigator — CHU de Clermont-Ferrand
Locations (1):
- CHU de Clermont-Ferrand, Clermont-Ferrand, Auvergne, France